CLINICAL TRIAL: NCT02119039
Title: Effect of CACICOL20 on Corneal Epithelial Healing After Cross-linking in Patients With Keratoconus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Katarzyna J. Witkowska, MD, PhD, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-070214
Record Dates: First submitted 2014-03-21; First posted 2014-04-21 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Keratoconus
Keywords: Cross-linking; RGTA OTR4120 (CACICOL20)
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- RGTA OTR 4120 (CACICOL20) (Experimental)
  Interventions: Device: RGTA OTR 4120 (CACICOL20)
- Genteal HA (Active Comparator)
  Interventions: Device: Genteal HA eye drops

INTERVENTIONS:
Device: RGTA OTR 4120 (CACICOL20)
  Arms: RGTA OTR 4120 (CACICOL20)
Device: Genteal HA eye drops
  Arms: Genteal HA

SUMMARY:
CACICOL20 is an ophthalmic solution based on the technology of RGTAs (ReGeneraTingAgents). It consists of large biopolymers, imitating the structure of heparansulphate. The protecting effect on different biological tissues and enhancement of wound healing has been described in several studies.

Keratoconus is a relatively common disease, with incidences ranging from 1.3 to 25 per 100,000 per year across different populations. Corneal collagen cross-linking represents a treatment option for these patients, aiming to prevent progression of the disease via stabilization of corneal microstructure. Corneal epithelial removal prior to the ultraviolet A/riboflavin cross-linking procedure significantly improves the outcome of the intervention, due to ameliorated distribution of riboflavin.

The aim of the present study is to investigate the effect of CACICOL20 on corneal epithelial wound closure after collagen cross-linking in patients with keratoconus. Results may lead to an improved management and pain reduction of patients with corneal epithelial defects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Presence of keratoconus
* Scheduled for corneal cross linking
* No ophthalmic surgery in the 3 months preceding the study

Exclusion Criteria:

* Participation in a clinical trial in the previous 3 weeks
* Topical use of aminoglycosid antibiotics
* Use of therapeutic or refractive contact lenses after surgery
* Known hypersensitivity to any component of the study medication or heparinoids or heparin
* Active ocular infection
* Presence of any abnormalities preventing reliable measurements as judged by the investigator
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to closure of the epithelial wound | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Bata AM, Witkowska KJ, Wozniak PA, Fondi K, Schmidinger G, Pircher N, Szegedi S, Aranha Dos Santos V, Pantalon A, Werkmeister RM, Garhofer G, Schmetterer L, Schmidl D. Effect of a Matrix Therapy Agent on Corneal Epithelial Healing After Standard Collagen Cross-linking in Patients With Keratoconus: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Oct 1;134(10):1169-1176. doi: 10.1001/jamaophthalmol.2016.3019. PMID 27584715